CLINICAL TRIAL: NCT01975701
Title: A Phase 2, Multicenter, Open-label Study of BGJ398 in Patients With Recurrent Resectable or Unresectable Glioblastoma
Brief Title: A Phase 2 Study of BGJ398 in Patients With Recurrent GBM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBGJ398X2201
Record Dates: First submitted 2013-10-28; First posted 2013-11-05 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Recurrent Glioblastoma or Other Glioma Subtypes
Keywords: BGJ398,; recurrent glioblastoma'; recurrent GBM,; FGFR,
MeSH Terms: conditions — Glioblastoma | interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BGJ398X (Experimental): To estimate anti-tumor efficacy of BGJ398
  Interventions: Drug: BGJ398

INTERVENTIONS:
Drug: BGJ398 — Capsule for oral use.

SUMMARY:
This is an open-label non-randomized, multicenter, phase II study of BGJ398 administered to adult patients with histologically confirmed GBM and/or other glioma subtypes with FGFR1-TACC1, FGFR3-TACC3 fusion and/or activating mutation in FGFR1, 2 or 3.

DETAILED DESCRIPTION:
Patients were enrolled in two groups. Group 1 enrolled patients who are not candidates for surgery. Group 2 was planned to enroll patients who are surgical candidates. Patients from both groups were evaluated for tumor response and progression by MRI every 8 weeks until disease progression or discontinuation from study using RANO criteria.

ELIGIBILITY:
Inclusion criteria:

1. Patients with histologically confirmed GBM and/or other glioma subtypes at the time of diagnosis or prior relapse.
2. Written documentation of local or central laboratory determination of amplification or translocation to FGFR1-TACC1, FGFR3-TACC-3 fusion and/or activating mutation in FGFR1, FGFR2,or FGFR3
3. RANO defined tumor progression by MRI in comparison to a prior scan
4. Patients must have received prior external beam radiotherapy and temozolomide.

Exclusion criteria:

1. History of another primary malignancy
2. Prior or current treatment with a FGFR inhibitor
3. Neurological symptoms related to underlying disease requiring increasing doses of corticosteroids
4. Patients must not be taking Enzyme Inducing Anti-Epileptic Drug (EIAED). If previously on an EIAED, the patient must be off of it for at least two weeks prior to study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-12-09 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (8):
  - Novartis Investigative Site, Los Angeles, California
  - University of California San Francisco Dept of Onc., San Francisco, California
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Novartis Investigative Site, Leuven, Belgium
- University Medical Center Utrecht, Utrecht, The Netherlands, Netherlands
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 26 patients included were enrolled in the non-Surgical group, and were treated with BGJ398 125 mg once daily in 28-day cycles, on a 3 weeks on/1 week off schedule (dosing days 1 to 21 of every 28-day cycle).
  No patients were enrolled in the surgical group.
Pre-assignment Details: Patients were planned to be enrolled in two groups:
  Group 1 (non-surgical group) targeted patients with response assessment in neuro-oncology (RANO) defined tumor progression not eligible for surgical resection.
  Group 2 (surgical group) targeted patients with recurrent disease eligible for cytoreductive surgery.
Groups:
- BGJ398X: 125 mg BGJ398 non surgical
Period: Overall Study
Arm/Group | BGJ398X
Started | 26
Completed | 1
Not Completed | 25
Not completed — Lost to Follow-up | 1
Not completed — Death | 23
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | BGJ398X
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  caucasian | 26

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: To assess the anti-tumor activity of BGJ398 for patients with GBM and/or other glioma subtypes that harbor FGFR1-TACC1, FGFR3-TACC3 fusion and/or activating mutation in FGFR1, 2 or 3 based on PFS6 (PFS rate at 6 months as defined by RANO criteria as assessed by the investigator)
Time Frame: 6 months
Population: full analysis set, patients censored
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BGJ398X
Number analyzed (Participants) | 24
months | 1.7 [1.05 to 2.80]

2. Secondary Outcome: Overall Response Rate
Description: To further assess the anti-tumor activity of BGJ398 for patients with GBM with an amplification, translocation, or activating mutation in FGFR1,2,3 or 4, based on Objective Response Rate (ORR - patients with measurable disease - as defined by RANO criteria as assessed by the investigator
Time Frame: 5 years
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BGJ398X
Number analyzed (Participants) | 26
Participants
  partial response | 2
  stable disease | 7
  progressive disease | 13
  unknown | 3
  missing | 1

3. Secondary Outcome: Overall Survival
Description: To further assess the anti-tumor activity of BGJ398 for patients with GBM and/or other glioma subtypes that harbor FGFR1-TACC1, FGFR3-TACC3 fusion and/or activating mutation in FGFR1, 2 and 3 based on Overall Survival
Time Frame: 5 years
Population: full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BGJ398X
Number analyzed (Participants) | 26
months | 6.74 [4.17 to 11.73]

4. Secondary Outcome: Safety and Tolerability
Description: Safety: type, frequency, and severity of AEs and SAEs; Tolerability: dose interruptions, reductions and dose intensity, and evaluations of laboratory values
Time Frame: 5 years
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BGJ398X
Number analyzed (Participants) | 26
Participants
  participants with dose interruptions | 13
  participants with dose reductions | 4

ADVERSE EVENTS:
Time Frame: All AEs reported in this record are treatment emergent AEs, collected from date of First Patient First Treatment until the completion of the safety follow-up ( 30 days after the Last Patient Last Treatment ) up to approximately 5 years.
Groups:
- Non Surg BGJ398 125 mg: Non Surg BGJ398 125 mg
Arm/Group | Non Surg BGJ398 125 mg
All-Cause Mortality (participants affected / at risk) | 3/26
Serious Adverse Events (participants affected / at risk) | 9/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non Surg BGJ398 125 mg (N=26)
Cataract (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Ataxia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Neurological decompensation (Nervous system disorders) | 2
Neurological symptom (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Cataract operation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non Surg BGJ398 125 mg (N=26)
Anaemia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Dry eye (Eye disorders) | 3
Eyelid ptosis (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 2
Fatigue (General disorders) | 9
Gait disturbance (General disorders) | 3
Mucosal inflammation (General disorders) | 2
Oedema peripheral (General disorders) | 3
Conjunctivitis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperlipasaemia (Metabolism and nutrition disorders) | 4
Hyperphosphataemia (Metabolism and nutrition disorders) | 20
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Aphasia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 6
Hemiparesis (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 4
Urinary incontinence (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
BGJ398 was out licensed and the indication was no longer pursued. Remaining patient continued treatment in post-trial settings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT01975701/SAP_000.pdf
  • Study Protocol (2015-04-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT01975701/Prot_001.pdf